CLINICAL TRIAL: NCT04148755
Title: The Accurateness of Endoscopic Ultrasound Elastography in the Guidance of EUS-FNA in Solid Pancreatic Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Mohamed Mahmoud, Assistant lecturer at internal medicine department, Assiut University
Other Study IDs: Elastography-FNA
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer
Keywords: EUS. Elastography, FNA
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elastography guided FNA: Those patients are going to have EUS elastography guided FNA
  Interventions: Procedure: Endoscopic ultrasound guided fine needle aspirate
- EUS. FNA: From records we are going to compare them with patients who had EUS without elastography guided FNA
  Interventions: Procedure: Endoscopic ultrasound guided fine needle aspirate

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided fine needle aspirate — All patients are going to have an EUS guided elastography with FNA of solid pancreatic lesions

SUMMARY:
To evaluate the role and effectiveness of EUS elastography as the guidance for direction of the site of fine needle aspirate (FNA) for tissue acquisition of solid pancreatic lesions

DETAILED DESCRIPTION:
Pancreatic cancer is one of the leading causes of cancer-related death. It has a poor 5-year survival rate of around8-9%. This is primarily because of most patients with pancreatic adenocarcinoma progress to either metastatic or locally advanced disease while in the asymptomatic phase. However, if pancreatic cancer is detected in the early stage (i.e., less than 2.0 cm), it has a relatively better prognosis.

Traditionally, transabdominal ultrasound or computed tomography CT scanning are used to diagnose pancreatic lesions. However, transabdominal ultrasound is limited because it cannot be used to visualize the entire pancreas due to intervening fat or air. Endoscopic ultrasonography (EUS) is currently an essential emerging tool for the work-up of pancreaticobiliary neoplasms. (EUS) is an ultrasound (US) technique in which the tip of the endoscope is equipped with a high-frequency transducer. High-resolution images of the pancreas can be obtained through the esophagus, stomach, and duodenum, without the disrupting effects of intervening gas, fat, and bone. EUS is now regarded as the most sensitive imaging modality for the detection of even a very small pancreatic lesion. Endoscopic ultrasound (EUS) elastography is a novel non-invasive technique that is used for the evaluation of pancreatic tissue which was first reported in 2006 and can be used for distinguishing benign from malignant pancreatic masses. Therefore, accurate detection of small cancers is important for reducing the mortality rate from pancreatic cancer. The equipment can be coupled with conventional EUS without the need for additional devices. There are two types of EUS elastography, strain and shear wave. Strain elastography estimates the stiffness and elasticity of the target tissue by measuring the degree of strain produced in response to compression. Shear wave elastography involves the emission of focused ultrasound from the probe to the target tissue, the so-called 'acoustic radiation force impulse' (ARFI), and the stiffness of the target tissue is then estimated by measuring the propagation speed of the shear wave. Only strain elastography is so far available for EUS. EUS elastography is used to characterize pancreatic masses and lymph node metastases of pancreatic cancer as well as to judge the severity of chronic pancreatitis with the evaluation of lesion elasticity EUS-guided fine needle aspiration (EUS-FNA) has been generally used for the sampling of pancreatic tissues since it was first reported in 1992. In general, 19G-25G caliber needles are inserted under EUS guidance for the pathological diagnosis of pancreatic cancer and lymph nodes and/or hepatic focal lesions. The overall complication rate of EUS-FNA is including complications such as pain, bleeding, and pancreatitis.

EUS FNA remains the gold standard in diagnosing pancreatic lesions and pancreatic cancer via tissue acquisition with a sensitivity of 80-85% and a specificity of 100 %, however, the diagnostic accuracy of EUS guided FNA is limited and EUS FNA can be associated with risks and complications. Many pre-procedural and procedural considerations must be assessed before performing EUS guided FNA. The location of the lesion, lack of adequate visualization, lack of experience of the endoscopist, lack of onsite pathology, and lack of adequate sampling are all limitations in diagnostic yield. False negatives can also occur in up to 40% of cases. In our multi-center experience, we are going to focus on the use of EUS elastography to direct the site of fine-needle aspiration in tissue acquisition of solid pancreatic lesions and its effect on the accuracy of diagnosis and detection of solid pancreatic lesions.

ELIGIBILITY:
Inclusion Criteria:

1 -All patients presented for EUS evaluation of solid pancreatic lesions 2-Accidentally discovered solid pancreatic lesions during EUS examination for any other cause

Exclusion Criteria:

1. Uncontrolled coagulopathy
2. Patients refused to enroll to the study.
3. Patients with cystic pancreatic lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are indicated for EUS evaluation of pancreatic lesions
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
The rate of Accurate diagnosis of pancreatic lesions | 2 years
The incidence and frequency of FNA passes | 2year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] McGuigan A, Kelly P, Turkington RC, Jones C, Coleman HG, McCain RS. Pancreatic cancer: A review of clinical diagnosis, epidemiology, treatment and outcomes. World J Gastroenterol. 2018 Nov 21;24(43):4846-4861. doi: 10.3748/wjg.v24.i43.4846. PMID 30487695
- [Background] Hara K, Yamao K, Mizuno N, Hijioka S, Sawaki A, Tajika M, Kawai H, Kondo S, Shimizu Y, Niwa Y. Interventional endoscopic ultrasonography for pancreatic cancer. World J Clin Oncol. 2011 Feb 10;2(2):108-14. doi: 10.5306/wjco.v2.i2.108. PMID 21603319
- [Background] Prado-Costa R, Rebelo J, Monteiro-Barroso J, Preto AS. Ultrasound elastography: compression elastography and shear-wave elastography in the assessment of tendon injury. Insights Imaging. 2018 Oct;9(5):791-814. doi: 10.1007/s13244-018-0642-1. Epub 2018 Aug 17. PMID 30120723
- [Background] Jani BS, Rzouq F, Saligram S, Lim D, Rastogi A, Bonino J, Olyaee M. Endoscopic Ultrasound-Guided Fine-Needle Aspiration of Pancreatic Lesions: A Systematic Review of Technical and Procedural Variables. N Am J Med Sci. 2016 Jan;8(1):1-11. doi: 10.4103/1947-2714.175185. PMID 27011940
- [Background] Jafri M, Sachdev AH, Khanna L, Gress FG. The Role of Real Time Endoscopic Ultrasound Guided Elastography for Targeting EUS-FNA of Suspicious Pancreatic Masses: A Review of the Literature and A Single Center Experience. JOP. 2016 Sep;17(5):516-524. PMID 28912670
- [Background] Weston BR, Bhutani MS. Optimizing Diagnostic Yield for EUS-Guided Sampling of Solid Pancreatic Lesions: A Technical Review. Gastroenterol Hepatol (N Y). 2013 Jun;9(6):352-63. PMID 23935542